CLINICAL TRIAL: NCT01092611
Title: Long-term Follow-up of Participants From Studies Evaluating the HIV Vaccine 732462
Brief Title: Long-term Follow-up of Participants From Studies Evaluating GSK HIV Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 114083; 2009-018097-64 (EudraCT Number)
Record Dates: First submitted 2010-03-22; First posted 2010-03-25 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: AIDS
Keywords: long-term follow-up study; HIV-infected subjects; HIV therapeutic vaccine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Blood Specimen Collection

ARMS (2):
- Group A (Other): Subjects who were administered the GSK HIV vaccine 732462 in primary studies and who accepted to participate in this study
  Interventions: Procedure: Blood collection; Biological: GSK HIV vaccine 732462
- Group B (Other): Subjects who were administered placebo in primary studies and who accepted to participate in this study
  Interventions: Procedure: Blood collection

INTERVENTIONS:
Procedure: Blood collection — Once a year after Visit 1 (during a maximum of 4 years). The samples will only be taken in conjunction with, and at the same time as, planned routine blood testing using the same needle-stick.
Biological: GSK HIV vaccine 732462 — No vaccine will be administered during this long-term follow-up study. Vaccines were administered during the primary studies.
  Arms: Group A

SUMMARY:
The purpose of this long-term follow-up study is to assess the long-term health status of HIV-infected subjects who previously participated in GSK-sponsored trials evaluating the investigational HIV vaccine 732462. This study will provide additional data concerning the long-term benefits/risks associated with vaccination.

No vaccine will be administered during the study period. Vaccines were administered during the primary studies.

DETAILED DESCRIPTION:
General information on the health of the subject and persistence of the cellular and humoral immune responses to study vaccination will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* HIV-infected subject.
* Previous participation in a study evaluating GSK HIV vaccine 732462.
* Written informed consent obtained from the subject.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If ANY exclusion criterion applies, the subject must not be included in the study:

• Subjects who did not receive a complete vaccination course in previous studies.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2010-03-22 (Actual); Primary Completion 2014-03-17 (Actual); Study Completion 2014-05-19 (Actual)

PRIMARY OUTCOMES:
Occurrence of Anti-Retroviral Therapy (ART) (re)-initiation or ART modification, and reason (for ART modification) | Once a year after Visit 1 (during a maximum of 4 years)
CD4 count | Once a year after Visit 1 (during a maximum of 4 years)
Viral load (VL) and method of measurement | Once a year after Visit 1 (during a maximum of 4 years)
Occurrence of HIV disease progression | Once a year after Visit 1 (during a maximum of 4 years)
Occurrence of each separate defining condition for HIV-disease progression | Once a year after Visit 1 (during a maximum of 4 years)
Occurrence of specific clinical events and death | Once a year after Visit 1 (during a maximum of 4 years)
Occurrence of adverse events (AEs) or serious adverse events (SAEs) considered by the Investigator to be related to vaccination (performed in the preceding vaccination study) | Once a year after Visit 1 (during a maximum of 4 years)
Occurrence of potential immune-mediated diseases (pIMDs) | Once a year after Visit 1 (during a maximum of 4 years)
Occurrence of SAEs related to study participation | Once a year after Visit 1 (during a maximum of 4 years)

SECONDARY OUTCOMES:
Time between dose 1 and ART (re)-initiation or ART modification | Once a year after Visit 1 (during a maximum of 4 years)
Time between dose 1 and CD4 count measurement | Once a year after Visit 1 (during a maximum of 4 years)
Time between dose 1 and VL measurement | Once a year after Visit 1 (during a maximum of 4 years)
Time between dose 1 and occurrence of HIV disease progression | Once a year after Visit 1 (during a maximum of 4 years)
Time between dose 1 and occurrence of each separate defining condition for HIV-disease progression | Once a year after Visit 1 (during a maximum of 4 years)
Antibody concentrations to vaccine antigens | Once a year after Visit 1 (during a maximum of 4 years)
Cell-mediated immunity responses | Once a year after Visit 1 (during a maximum of 4 years)
Additional exploratory immunogenicity endpoints (other T-cell immune markers or T-cell functional assays) | Once a year after Visit 1 (during a maximum of 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (27):
- United States (10):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Annandale, Virginia
  - GSK Investigational Site, Seattle, Washington
- France (4):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
- Germany (8):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Spain (5):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles, Madrid
  - GSK Investigational Site, Valencia

REFERENCES:
- [Derived] Harrer T, Dinges W, Roman F; TH-HIV-011 study group. Long-term follow-up of HIV-1-infected adults who received the F4/AS01B HIV-1 vaccine candidate in two randomised controlled trials. Vaccine. 2018 May 3;36(19):2683-2686. doi: 10.1016/j.vaccine.2018.03.043. Epub 2018 Mar 30. PMID 29606517
- See also: Results for study 114083 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/114083?search=study&b%22b''%22#rs